CLINICAL TRIAL: NCT02351115
Title: Assessment of Staccato® Alprazolam on the EEG Photoparoxysmal Response in Patients With Epilepsy
Brief Title: Staccato Alprazolam and Photoparoxysmal Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: The Epilepsy Study Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-002-202
Record Dates: First submitted 2015-01-19; First posted 2015-01-30 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sequence BEADC (Experimental): A=Placebo, B=Inhaled Alprazolam 0.5 mg, C=Inhaled Alprazolam 1 mg, D= Inhaled Alprazolam 2 mg, E=Placebo
  Interventions: Drug: A=Placebo; Drug: B=Inhaled Alprazolam 0.5 mg; Drug: C=Inhaled Alprazolam 1 m; Drug: D= Inhaled Alprazolam 2 mg; Drug: E=Placebo
- Sequence CDAEB (Experimental): A=Placebo, B=Inhaled Alprazolam 0.5 mg, C=Inhaled Alprazolam 1 mg, D= Inhaled Alprazolam 2 mg, E=Placebo
  Interventions: Drug: A=Placebo; Drug: B=Inhaled Alprazolam 0.5 mg; Drug: C=Inhaled Alprazolam 1 m; Drug: D= Inhaled Alprazolam 2 mg; Drug: E=Placebo
- Sequence DEBAC (Experimental): A=Placebo, B=Inhaled Alprazolam 0.5 mg, C=Inhaled Alprazolam 1 mg, D= Inhaled Alprazolam 2 mg, E=Placebo
  Interventions: Drug: A=Placebo; Drug: B=Inhaled Alprazolam 0.5 mg; Drug: C=Inhaled Alprazolam 1 m; Drug: D= Inhaled Alprazolam 2 mg; Drug: E=Placebo
- Sequence EDBAC (Experimental): A=Placebo, B=Inhaled Alprazolam 0.5 mg, C=Inhaled Alprazolam 1 mg, D= Inhaled Alprazolam 2 mg, E=Placebo
  Interventions: Drug: A=Placebo; Drug: B=Inhaled Alprazolam 0.5 mg; Drug: C=Inhaled Alprazolam 1 m; Drug: D= Inhaled Alprazolam 2 mg; Drug: E=Placebo
- Sequence CABED (Experimental): A=Placebo, B=Inhaled Alprazolam 0.5 mg, C=Inhaled Alprazolam 1 mg, D= Inhaled Alprazolam 2 mg, E=Placebo
  Interventions: Drug: A=Placebo; Drug: B=Inhaled Alprazolam 0.5 mg; Drug: C=Inhaled Alprazolam 1 m; Drug: D= Inhaled Alprazolam 2 mg; Drug: E=Placebo

INTERVENTIONS:
Drug: A=Placebo
Drug: B=Inhaled Alprazolam 0.5 mg
Drug: C=Inhaled Alprazolam 1 m
Drug: D= Inhaled Alprazolam 2 mg
Drug: E=Placebo

SUMMARY:
The purpose of this study is to determine whether people who usually have photosensitive epilepsy will show a reduction in epileptic activity when they take a single dose of Staccato Alprazolam as compared to placebo.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether people who usually have photosensitive epilepsy will show a reduction in epileptic activity when they take a single dose of Staccato Alprazolam as compared to placebo. People with photosensitive epilepsy have changes on their electroencephalogram (EEG) when shown flashing lights. Three dose levels of Staccato Alprazolam will be compared to placebo.

This study will also assess the level of sedation of Staccato Alprazolam compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 60 years, inclusive
* Body mass index (BMI) ≥18 and ≤35 kg/m2
* Able to speak, read, and understand English and willing and able to provide written informed consent on an IRB-approved form before the initiation of any study procedures
* A diagnosis and history of a photoparoxysmal response on EEG with or without a diagnosis of epilepsy for which patients are on 0-2 concomitant antiepileptic drugs
* At least 3 of the EEGs performed during the screen visit must have a reproducible IPS-induced photoparoxysmal response (PPR) on EEG of at least 3 points on a frequency assessment scale in at least one eye condition
* In otherwise good general health as determined by a complete medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, and urinalysis
* Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method throughout the study and for 1 week following the end of the study. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone

Exclusion Criteria:

* History of non-epileptic seizures (e.g. metabolic, structural, or pseudo-seizures)
* History of seizure worsening in response to narrow spectrum drugs
* An active CNS infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results
* Use of more than 2 concomitant AEDs for epilepsy treatment
* Subjects taking known inhibitors or inducers of CYP3A , including carbamazepine
* Subjects with a history of allergic reactions to alprazolam or other benzodiazepines
* Treatment with an investigational drug within 30 days (or within 5 half-lives of the investigational drug, if >30 days) before Visit 2
* A history within the past 1 year of drug or alcohol dependence or abuse
* Positive urine screen for drugs of abuse at Visit 1 - Screening
* A history of HIV-positivity
* Female subjects who have a positive pregnancy test at screening or prior to test sessions or are breastfeeding
* History of acute narrow angle glaucoma, Parkinson's disease, hydrocephalus, or history of significant head trauma
* Subjects who have a current history of asthma, chronic obstructive lung disease (COPD), or any lung disease associated with bronchospasm
* Subjects who use medications to treat airways disease, such as asthma or COPD
* Subjects who have any acute respiratory signs/symptoms (e.g., wheezing)
* Clinically significant ECG abnormality including (but not limited to) any of the following conduction abnormalities or dysrhythmias: atrial fibrillation, mean QTcF (QT interval corrected for heart rate using Fridericia's method) interval >450 msec, ventricular rate <45 beats/min, second or third degree AV block, left bundle branch block, or evidence of prior myocardial infarction (MI) or acute ischemia
* Hypotension (systolic blood pressure ≤90 mm Hg, diastolic blood pressure ≤50 mm Hg), or hypertension (systolic blood pressure ≥140 mm Hg, diastolic blood pressure ≥100 mm Hg) measured while seated at screening or baseline
* Significant hepatic, renal, gastroenterologic, cardiovascular (including ischemic heart disease and congestive heart failure), endocrine, neurologic (including history of seizures or stroke), or hematologic disease
* Any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Isojarvi, MD, Study Chair — Engage Therapeutics, Inc.
Locations (3):
- United States (3):
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - New York University Epilepsy Center, New York, New York
  - University of Pennsylvania - Penn Epilepsy Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 10 days of request approval
Access Criteria: Approval of formal request for access
URL: http://alexza.com

RESULTS

PARTICIPANT FLOW:
Groups:
- BEADC: Patient receiving treatment sequence BEADC
- CDAEB: Patient receiving treatment sequence CDAEB
- DEBAC: Patient receiving treatment sequence DEBAC
- EDBAC: Patient receiving treatment sequence EDBAC
- CABED: Patient receiving treatment sequence CABED
Period: Overall Study
Arm/Group | BEADC | CDAEB | DEBAC | EDBAC | CABED
Started | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects treated
Groups:
- BEADC BEADC: Patient receiving treatment sequence BEADC
- Total: Total of all reporting groups
Arm/Group | BEADC BEADC | CDAEB | DEBAC | EDBAC | CABED | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (0) | 23 (0) | 27 (0) | 39 (0) | 23 (0) | 27.2 (6.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 5
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Ethnicity: Not Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 4
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
  Race: Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Race: Not Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 4
  Race: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Change From Pretreatment Baseline in the Standardized Photosensitivity Range (SPR)
Description: Photosensitivity describes the presentation of an epileptiform EEG response (photoparoxysmal response) from exposure to intermittent photic stimulation (IPS). SPR is the number of frequency steps (2, 5, 8, 10, 13, 15, 18, 20, 23, 25, 30, 40, 50 and 60 Hz). between the upper and lower limits of sensitivity to IPS for that patient at that time, in order not to evoke seizures. Thus a reduction (-change) means the intervention is working (desired effect on sensitivity)
Time Frame: SPR was recorded pretreatment, 2, 10, 30 min, 1, 2, 4, and 6 hr post each study drug administration The maximum change from baseline occurred at: 10 min for alprazolam 2 mg, 1 hour for alprazolam 0.5 and 1 mg and placebo
Population: All 5 patients received all 4 treatments (crossover design)
Measure: Mean (90% Confidence Interval); unit: Number of frequency steps
Groups:
- Inhaled Placebo: All patients receiving inhaled placebo in this 4 treatment complete crossover study
- Staccato Alprazolam, 0.5 mg: All patients receiving 0.5 mg inhaled alprazolam in this 4 treatment complete crossover study
- Staccato Alprazolam, 1 mg: All patients receiving 1 mg inhaled alprazolam in this 4 treatment complete crossover study
- Staccato Alprazolam, 2 mg: All patients receiving 2 mg inhaled alprazolam in this 4 treatment complete crossover study
Arm/Group | Inhaled Placebo | Staccato Alprazolam, 0.5 mg | Staccato Alprazolam, 1 mg | Staccato Alprazolam, 2 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
Number of frequency steps | -0.2 [-1.87 to 1.47] | -4.4 [-6.98 to -1.82] | -5.2 [-7.85 to -2.55] | -4.8 [-7.99 to -1.61]

2. Secondary Outcome: Maximum Sedation Using Visual Analog Scale (Sedated-Alert)
Description: Maximum change (in mm) from pretreatment baseline in level of sedation reported by the patient on a 100 mm line anchored by Sedated (0) and Alert (100)
Time Frame: Sedation was recorded pretreatment, 2, 10, 30 min, 1, 2, 4, and 6 hr post each study drug administration The maximum change from baseline occurred at:: 30 min for alprazolam 1 mg, 1 hour for alprazolam 0.5 and 2 mg, and 4 hours for placebo
Population: All 5 patients received each of the 4 treatments after washout (crossover design)
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Inhaled Placebo | Staccato Alprazolam, 0.5 mg | Staccato Alprazolam, 1 mg | Staccato Alprazolam, 2 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | -5.3 [-23.84 to 13.34] | -58 [-82.77 to -33.23] | -67.4 [-87.47 to -47.33] | -70.6 [-94.06 to -47.14]

3. Secondary Outcome: Maximum Sedation Using Visual Analog Scale (Sleepy-Awake)
Description: Maximum change (in mm) from pretreatment baseline in level of sedation reported by each subject on a 100 mm line anchored by Sleepy (0) and Awake (100)
Time Frame: Sleepiness was recorded pretreatment, 2, 10, 30 min, 1, 2, 4, and 6 hr post each study drug administration The maximum change from baseline occurred: at: 30 min for alprazolam 1 mg, 1 hour for alprazolam 0.5 and 2 mg and placebo
Population: All 5 patients received each of the 4 treatments after washout (crossover design)
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Inhaled Placebo | Staccato Alprazolam, 0.5 mg | Staccato Alprazolam, 1 mg | Staccato Alprazolam, 2 mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
units on a scale | -9.2 [-26.33 to 7.93] | -54 [-72.59 to -35.31] | -58.8 [-76.01 to -41.59] | -58.8 [-69.4 to -48.2]

4. Secondary Outcome: Correlation of Plasma Concentrations of Alprazolam With Pharmacodynamic Effects on Standardized Photosensitivity Range (SPR)
Description: Pearson correlation of all paired plasma concentrations of alprazolam (PK) with pharmacodynamic effect on SPR (PD) for each alprazolam dose
Time Frame: Pretreatment, 2, 10, 30 min, 1, 2, 4, and 6 hr post each study drug administration
Population: PK-PD population pairs, All 5 crossover subjects by alprazolam treatment received
  Number of PK-PD pairs per dose (n) = 35 (7 time points x 5 subjects)
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Staccato Alprazolam, 0.5 mg | Staccato Alprazolam, 1 mg | Staccato Alprazolam, 2 mg
Number analyzed (Participants) | 5 | 5 | 5
correlation coefficient | -0.454 (0.206) | -0.534 (0.286) | -0.410 (0.168)

5. Secondary Outcome: Correlation of Plasma Concentrations of Alprazolam With Pharmacodynamic Effects on Visual Analog Scale (Sedated-Alert)
Description: Pearson correlation of all paired plasma concentrations of alprazolam (PK) with pharmacodynamic effect on Sedation (PD) for each alprazolam dose
Time Frame: Pretreatment, 2, 10, 30 min, 1, 2, 4, and 6 hr post each study drug administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Staccato Alprazolam, 0.5 mg | Staccato Alprazolam, 1 mg | Staccato Alprazolam, 2 mg
Number analyzed (Participants) | 5 | 5 | 5
correlation coefficient | -0.350 (0.122) | -0.567 (0.322) | -0.623 (0.388)

6. Secondary Outcome: Correlation of Plasma Concentrations of Alprazolam With Pharmacodynamic Effects on Visual Analog Scale (Sleepy-Awake)
Description: Pearson correlation of all paired plasma concentrations of alprazolam (PK) with pharmacodynamic effect on Sleepiness (PD) for each alprazolam dose
Time Frame: Pretreatment, 2, 10, 30 min, 1, 2, 4, and 6 hr post each study drug administration
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Staccato Alprazolam, 0.5 mg | Staccato Alprazolam, 1 mg | Staccato Alprazolam, 2 mg
Number analyzed (Participants) | 5 | 5 | 5
correlation coefficient | -0.449 (0.201) | -0.582 (0.339) | -0.586 (0.343)

ADVERSE EVENTS:
Time Frame: Each subject was questioned about adverse events (AEs) at 2 min, 10 min, 30 min, 1 hr, 2 hr, 4 hr, and 6 hr post study drug administration for each study drug.
Groups:
- Staccato® Alprazolam, 0.5 mg: All patients receiving 0.5 mg inhaled alprazolam in this 4 treatment complete crossover study
- Staccato® Alprazolam, 1 mg: All patients receiving 1 mg inhaled alprazolam in this 4 treatment complete crossover study
- Staccato® Alprazolam, 2 mg: All patients receiving 2 mg inhaled alprazolam in this 4 treatment complete crossover study
Arm/Group | Inhaled Placebo | Staccato® Alprazolam, 0.5 mg | Staccato® Alprazolam, 1 mg | Staccato® Alprazolam, 2 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5 | 3/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=5) | Staccato® Alprazolam, 0.5 mg (N=5) | Staccato® Alprazolam, 1 mg (N=5) | Staccato® Alprazolam, 2 mg (N=5)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No